CLINICAL TRIAL: NCT04931017
Title: Metformin for Chemoprevention of Lung Cancer in High-Risk Overweight or Obese Individuals
Brief Title: Metformin for Chemoprevention of Lung Cancer in Overweight or Obese Individuals at High Risk for Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2021-06112; NCI-2021-06112 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI20-04-01 (Other: Northwestern University); NWU20-04-01 (Other: DCP); P30CA060553 (NIH); UG1CA242643 (NIH)
Record Dates: First submitted 2021-06-17; First posted 2021-06-18 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — Biopsy; Specimen Handling; Bronchoscopy; Metformin

STUDY DESIGN:
Intervention Model Description: This is a partial crossover model whereby the no-treatment subjects will receive the drug after being controls.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A - Former Smokers (metformin ER) (Experimental): Participants receive metformin ER PO QD for 26 weeks in the absence of unacceptable toxicity. Participants undergo bronchoscopy biopsy and blood sample collection at screening, and week 13.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Bronchoscopy; Drug: Extended Release Metformin Hydrochloride; Other: Questionnaire Administration
- Cohort B - Former Smokers (metformin ER with waiting period) (Active Comparator): Participants receive no intervention for 26 weeks, then cross-over to Cohort A. Participants undergo bronchoscopy biopsy and blood sample collection at screening, at week 26, and at 13 weeks after cross-over to Cohort A.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Bronchoscopy; Drug: Extended Release Metformin Hydrochloride; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bronchoscopy — Undergo bronchoscopy
Drug: Extended Release Metformin Hydrochloride — Given PO
  Other Names: ER Metformin Hydrochloride; Extended-release Metformin Hydrochloride; Glucophage XR; Glumetza; Metformin Hydrochloride Extended Release
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial determines the effect of metformin extended release on the risk for developing lung cancer in overweight/obese patients that are at high-risk for developing lung cancer. Metformin is widely used to treat type II diabetes and has a long history of safety and minimal side effects. At similar dosage, the drug may have potential anti-cancer activity. Metformin use has been associated with improved survival in patients with non-small cell lung carcinoma, a specific type of lung cancer, and it has also been shown to enhance immune mobilization against tumors. This trial aims to see whether metformin extended release as a preventative treatment may lower the chance of developing lung cancer, and whether it may help patients' immune system learn ("reprogram") to lower a certain type of immune cell (called regulatory T cells) that are linked to tumor development.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the effect of metformin treatment on the expression of programmed cell death protein 1 (PD-1) on airway regulatory T cells (Tregs) in overweight and obese individuals at high risk for lung cancer.

SECONDARY OBJECTIVES:

I. Estimated PD-1 expression of pulmonary Tregs change in Cohort B during the wait period (26 weeks with no treatment).

II. To examine the impact of metformin on circulating immune cell subsets of blood.

III. To evaluate the effect of metformin treatment on the expression of PD-1 on airway regulatory T cells (Tregs) in overweight and obese current smokers at high risk for lung cancer

EXPLORATORY OBJECTIVES:

I. To examine the impact of metformin on cancer-related transcriptome features of airway lesions.

II. To examine the impact of metformin on immune profile of pulmonary parenchyma represented by bronchoalveolar lavage (BAL).

III To examine the impact of metformin on histologic progression of abnormal airway lesions.

IV. To examine the impact of metformin on serum adipokines and inflammatory cytokines.

OUTLINE: Participants are randomized to 1 of 2 cohorts.

COHORT A: Former Smokers - Participants receive metformin extended release (ER) orally (PO) once daily (QD) for 26 weeks in the absence of unacceptable toxicity. Participants undergo bronchoscopy biopsy and blood sample collection at screening, and week 13.

COHORT B: Former Smokers - Participants receive no intervention for 26 weeks, then cross-over to cohort A. Participants undergo bronchoscopy biopsy and blood sample collection at screening, at week 26, and at 13 weeks after cross-over to Cohort A.

COHORT C: Current Smokers - Participants receive metformin extended release (ER) orally (PO) once daily (QD) for 26 weeks in the absence of unacceptable toxicity. Participants undergo bronchoscopy biopsy and blood sample collection at screening, and week 13.

After completion of study treatment, participants are followed up at weeks 30-32 (Cohorts A and C) and weeks 56-58 (Cohort B).

ELIGIBILITY:
Inclusion Criteria:

* Former smokers (male and female) with a >= 20 pack year smoking history
* Quit smoking >= 12 months prior to enrollment
* Prostate, Lung, Colorectal and Ovarian Cancer Screening Trial (PLCOm2012) Lung Cancer Risk Prediction Score > 1.34%
* Overweight

  * Body mass index (BMI) > 25 and
  * Waist circumference

    * Female > 88 cm (35")
    * Male > 102 cm (40")
* Age greater than 30 years. Participants younger than 30 years are unlikely to accrue enough smoking exposure followed by enough time after quitting (>12 months) to qualify
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Leukocytes >= 3,000/microliter
* Absolute neutrophil count (ANC) >= 1,000/microliter
* Platelets >= 100,000/microliter
* Total bilirubin =< 1.5 x institutional upper limit of normal (IULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 x IULN
* Estimated glomerular filtration rate (eGFR) > 45 ml/min/1.73 m^2 (eGFR will be calculated using the equation Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] creatinine)
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured
* Patients on chronic suppressive antiviral therapy for herpes simplex virus (HSV) are eligible
* The effects of metformin ER on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Current or previous diagnosis of diabetes mellitus (type I or type II diabetes)
* Use of metformin within the past 2 years
* Use of GLP-1 agonists within 6 weeks prior to enrollment
* Glycosylated hemoglobin A1C (HbA1c) > 8%
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to metformin ER
* Participants currently using immunosuppressive medication, including systemic steroids (not inhalational) and episodic use of inhaled steroids are excluded from this trial due to the potential impact of these treatments on the primary trial endpoint
* Participants receiving any other investigational agents
* History of chronic alcohol use or abuse defined by any one of the following:

  * Average consumption of 3 or more alcohol containing beverages daily in the past 12 months
  * Consumption of 7 or more alcoholic beverages within a 24 hour period in the past 12 months
* Acute or chronic liver disease, evidence of hepatitis (infectious or autoimmune), cirrhosis or portal hypertension
* History of or current condition predisposing to increased risk for lactic acidosis such as: severe congestive heart failure (New York Heart Association [NYHA] class III or IV), metabolic acidosis, severe liver disease, or renal failure
* Uncontrolled intercurrent illness or psychiatric illness/social situations that would or limit compliance with study requirements
* Pregnant women are excluded from this study. Metformin ER is a class B agent that was not teratogenic in rats and rabbits at doses representing 3 and 6 times the maximum recommended human daily dose of 2000 mg; however, animal reproduction studies are not always predictive of human response. Because there is an unknown but potential risk for adverse events (AEs) in nursing infants secondary to treatment of the mother with metformin ER, breastfeeding should be discontinued if the mother is treated with metformin ER
* Biopsy with invasive carcinoma of the lung or carcinoma in situ

  * Participants with prior stage 1 non-small cell lung cancer (NSCLC) diagnosis are allowed to participate, as long as there has been 12 months since the completion of cancer treatment prior to enrollment with no evidence of recurrence or second primary cancer

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
PD-1 expression of pulmonary regulatory T cells (Tregs) before and after metformin extended release (ER) treatment | Pre- to post-treatment
  Change from pre- to post-metformin extended release (ER) treatment in cell surface PD-1 expression levels of pulmonary (BAL) Tregs, measured as mean fluorescent intensity (MFI). Changes in MFI due to metformin ER treatment among all n = 40 subjects will be used for the primary analysis.

SECONDARY OUTCOMES:
Estimated PD-1 expression of pulmonary Tregs change in cohort B during the wait period (6 months with no treatment) | Randomization to week 26
  This is the estimate of change in MFI following the 6-month wait period among n = 20 subjects randomized to the wait-list arm. This will confirm the stability of the PD-1 expression of pulmonary Tregs over time.
Circulating immune cells | Pre- to post-treatment
  Circulating immune cell composition between blood samples collected pre- and post-metformin ER treatment to assess the effect of metformin ER on circulating immune cells and to identify potential biomarkers of metformin ER response.

OTHER OUTCOMES:
Airway gene expression | Up to study completion
  RNA sequencing of endobronchial biopsies will be performed at visually normal mainstem airway for each participant. The analysis of the RNA seq data will be an unsupervised comparison of differentially expressed genes with and without metformin ER exposure.
Examination of the immune profile of pulmonary parenchyma represented by bronchoalveolar lavage | Pre- to post-treatment
  This will compare the immune composition of bronchoalveolar lavage samples of participants before and after metformin exposure. Specifically, the prevalence and composition of myeloid derived suppressor cells (MDSCs) as well as monocyte, macrophage and dendritic cells will be assessed.
Histologic progression | Up to study completion
  Bronchoscopic biopsies of at least 6 standard sites will be graded on the World Health Organization (WHO) scale of dysplasia and assigned numerical scores from 1 (normal) to 8 (invasive cancer). Each lesion will be classified as complete response (CR), partial response (PR), stable disease (SD) or progressive disease (PD) and each response rate will be calculated on a per-site and a per-participant basis. Additional measures of dysplasia will include the average dysplastic score and the dysplasia index (% of sites with dysplasia score >= 3 (mild dysplasia)). Changes in maximum dysplasia will be analyzed using a paired t test to determine whether a reduction occurs.
Examination of the effect of metformin on systemic adipokines and inflammatory cytokines | Pre- to post-treatment
  Frozen sera will be analyzed by commercial enzyme-linked immunosorbent assay kits for levels of leptin, adiponectin, resistin, IL6 and TNFalpha. Pre- and post-treatment serum levels will be compared in parametric paired testing.

CONTACTS AND LOCATIONS:
Overall Officials: Saikrishna S Yendamuri, Principal Investigator — Roswell Park University
Locations (4):
- United States (2):
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - Roswell Park Cancer Institute, Buffalo, New York
- Canada (2):
  - BC Cancer Research Centre, Vancouver, British Columbia
  - University of British Columbia Hospital, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm